CLINICAL TRIAL: NCT06303804
Title: Prevention of Opioid Misuse and Overdose Deaths Among Hispanic/Latinx Adolescents: A Family-based Perspective
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Alejandra Fernandez, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0837
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Opioid Misuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational videos arm (Experimental)
  Interventions: Behavioral: Educational videos

INTERVENTIONS:
Behavioral: Educational videos — Participants will be delivered a link to complete demographic information and the initial assessment. Upon completing the (initial) pre-test knowledge assessment, participants will be sent links to the three educational videos staggered across 7 days. Educational videos will determine gaps in knowledge related to opioid use and overdose based on questionnaire responses. Upon the completion of the 7 days, participants will be sent a link to the (final) post-test knowledge assessment to complete.

SUMMARY:
The purpose of this study is to develop culturally-competent family-focused educational modules targeting opioid knowledge and attitudes (including targeting safe storage and prevention of accidental opioid overdose in adolescent populations) and examine changes acceptability, knowledge, and attitudes scores

ELIGIBILITY:
Inclusion Criteria:

* Must identify as Hispanic/Latino/a descent
* Have an adolescent between the ages of 15 and 17 years old living in their home a majority of the time
* Have English or Spanish proficiency

Exclusion Criteria:

* Adolescent or parent currently in opioid treatment
* Parent self-reports a substance use (including opioid use) disorder for themselves or adolescent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the educational materials presented via the educational videos, including cultural congruence as assessed by a questionnaire | end of study (Day 7)
  This questionnaire has 10 questions that is measured on a Likert scale from 1-4, higher number indicating more acceptability.
Changes in opioid related knowledge as assessed by a questionnaire | Baseline, end of study (Day 7)
  This has 3 subscales
  1. Brief Opioid Overdose Knowledge (BOOK)
     This has 12 questions and each is scored from 0(true), 1(false) for a maximum score of 12, higher score indicating more knowledge
  2. Opioid Overdose Knowledge Scale (OOKS)
     This has 9 questions, and participants have to identify all correct answers. Score ranges from 0(no correct answers) -33 (identified all correct answers) higher score indicates more knowledge
  3. Opioid Overdose Attitude Scale (OOAS)
  This has 28 questions scored on a Likert scale from 1(completely disagree)-5(completely agree), higher number indicating more positive attitude

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Fernandez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No